CLINICAL TRIAL: NCT03479307
Title: A Multi-Center, Double-Masked, Randomized, Vehicle- and Active-Controlled, Phase 3 Study Evaluating the Efficacy and Safety of Bilastine Ophthalmic Solution 0.6% Compared to Vehicle and Zaditen (Ketotifen Ophthalmic Solution 0.025%) for the Treatment of Allergic Conjunctivitis in the Conjunctival Allergen Challenge (Ora-CAC®) Model
Brief Title: A Study Evaluating Bilastine Ophthalmic Solution 0.6% in the Conjunctival Allergen Challenge (Ora-CAC®) Model.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BOFT-0218/AC-CAC
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2021-11

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Ketotifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bilastine Ophthalmic Solution 0.6% (Experimental): Bilastine Ophthalmic Solution 0.6%
  1 drop in each eye at 2 separate times during an 8 day period.
  Interventions: Drug: Bilastine Ophthalmic Solution 0.6%
- Ketotifen Ophthalmic Solution 0.025% (Zaditen) (Active Comparator): Ketotifen Ophthalmic Solution 0.025% (Zaditen)
  1 drop in each eye at 2 separate times during an 8 day period.
  Interventions: Drug: Ketotifen Ophthalmic Solution 0.025% (Zaditen)
- Vehicle of Bilastine Ophthalmic Solution (Placebo Comparator): Vehicle of Bilastine Ophthalmic Solution
  1 drop in each eye at 2 separate times during an 8 day period.
  Interventions: Drug: Vehicle of Bilastine Ophthalmic Solution

INTERVENTIONS:
Drug: Bilastine Ophthalmic Solution 0.6% — 1 drop in each eye at 2 separate times during an 8 day period.
  Arms: Bilastine Ophthalmic Solution 0.6%
Drug: Ketotifen Ophthalmic Solution 0.025% (Zaditen) — 1 drop in each eye at 2 separate times during an 8 day period.
  Other Names: Zaditen
  Arms: Ketotifen Ophthalmic Solution 0.025% (Zaditen)
Drug: Vehicle of Bilastine Ophthalmic Solution — 1 drop in each eye at 2 separate times during an 8 day period.
  Arms: Vehicle of Bilastine Ophthalmic Solution

SUMMARY:
To evaluate the efficacy of Bilastine ophthalmic solution 0.6% compared to vehicle and Zaditen (Ketotifen ophthalmic solution 0.025%) for the treatment of the signs and symptoms of allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years old
* be willing and able to avoid all disallowed medications and contact lenses
* must have a pregnancy test if of childbearing potential
* must be able to read an eye chart from 10 feet away

Exclusion Criteria:

* must not have any allergies to the study medications
* must not have any ocular or non ocular condition that investigator feels will interfere with study parameters
* must not have used immunotherapy in the last 2 years
* must not have used an investigational drug or device in the past 30 days or concurrently enrolled in another investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Cornea Consultants of AZ, Phoenix, Arizona
  - East West Eye Institute, Torrance, California
  - Andover Eye Associates, Andover, Massachusetts
  - Apex Eye, Mason, Ohio
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - Total Eye Care, P.A., Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomes PJ, Ciolino JB, Arranz P, Hernandez G, Fernandez N. Bilastine 0.6% Preservative-free Eye Drops: A Once-daily Treatment for Allergic Conjunctivitis. J Investig Allergol Clin Immunol. 2024 Jun 17;34(3):167-176. doi: 10.18176/jiaci.0894. Epub 2023 Feb 23. PMID 36811846

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bilastine Ophthalmic Solution 0.6% | Ketotifen Ophthalmic Solution 0.025% (Zaditen) | Vehicle of Bilastine Ophthalmic Solution
Started | 91 | 90 | 47
Completed | 90 | 89 | 47
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilastine Ophthalmic Solution 0.6% | Ketotifen Ophthalmic Solution 0.025% (Zaditen) | Vehicle of Bilastine Ophthalmic Solution | Total
Number analyzed (Participants) | 91 | 90 | 47 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 85 | 89 | 43 | 217
  >=65 years | 6 | 1 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (12.88) | 41.7 (12.1) | 45.1 (16.03) | 44.1 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 53 | 25 | 136
  Male | 33 | 37 | 22 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 6 | 27
  Not Hispanic or Latino | 80 | 79 | 41 | 200
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 14 | 13 | 6 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 25 | 27 | 14 | 66
  White | 49 | 48 | 26 | 123
  More than one race | 2 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 91 | 90 | 47 | 228
Ocular Itching- Baseline [Mean (Standard Deviation); unit: units on a scale] — The primary efficacy measure was ocular itching evaluated by the subject at 3 (± 1), 5 (±1), and 7 (± 1) minutes post-CAC (Conjunctival Allergen Challenge) at Visit 4b (Day 1: 16h post-treatment) and Visit 5 (Day 8 ±3, 15 minutes post-treatment), using a 0 to 4 Ora Calibra scale (0 = None , 4= An incapacitating itch with an irresistible urge to rub).
  The baseline measures for this primary outcome will be the "pre-CAC" values (Pre-Conjunctival Allergen Challenge).
  units on a scale
    Visit 4b: Pre-CAC | 0.014 (0.0945) | 0.011 (0.1054) | 0.043 (0.2949) | 0.023 (0.1649)
    Visit 5: Pre-CAC | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: The primary efficacy measure was ocular itching evaluated by the subject at 3 (± 1), 5 (±1), and 7 (± 1) minutes post-CAC (Conjunctival Allergen Challenge) at Visits 4b and 5, using a 0 to 4 Ora Calibra scale (0 = None , 4= An incapacitating itch with an irresistible urge to rub).
Time Frame: The outcome measure was assessed at Visit 4b (Day 1: 16h post-treatment) and Visit 5 (Day 8 ±3, 15 minutes post-treatment).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bilastine Ophthalmic Solution 0.6% | Ketotifen Ophthalmic Solution 0.025% (Zaditen) | Vehicle of Bilastine Ophthalmic Solution
Number analyzed (Participants) | 91 | 90 | 47
units on a scale
  Visit 4b: 3 minutes Post- CAC | 1.609 (0.9013) | 1.886 (0.9504) | 2.219 (0.9644)
  Visit 4b: 5 minutes Post- CAC | 1.750 (0.9508) | 1.919 (0.9670) | 2.490 (0.8996)
  Visit 4b: 7 minutes Post- CAC | 1.747 (1.0283) | 1.894 (0.9606) | 2.526 (0.9035)
  Visit 5: 3 minutes Post- CAC | 0.669 (0.7926) | 0.658 (0.6745) | 1.840 (0.9258)
  Visit 5: 5 minutes Post- CAC | 0.828 (0.8879) | 0.902 (0.8208) | 2.011 (0.9058)
  Visit 5: 7 minutes Post- CAC | 0.826 (0.8901) | 0.981 (0.9224) | 1.931 (0.8703)
Statistical Analysis 1: Comparison: Bilastine Ophthalmic Solution 0.6% vs Vehicle of Bilastine Ophthalmic Solution; Treatment Difference (95% CI): Bilastine Ophthalmic Solution 0.6% arm minus Vehicle of Bilastine Ophthalmic Solution arm at Visit 4b (including all time points); Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.710, 95% CI 2-sided [-1.013 to -0.407]
Statistical Analysis 2: Comparison: Bilastine Ophthalmic Solution 0.6% vs Vehicle of Bilastine Ophthalmic Solution; Treatment Difference (95% CI): Bilastine Ophthalmic Solution 0.6% arm minus Vehicle of Bilastine Ophthalmic Solution arm at Visit 5 (including all time points); Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.167, 95% CI 2-sided [-1.439 to -0.895]
Statistical Analysis 3: Comparison: Ketotifen Ophthalmic Solution 0.025% (Zaditen) vs Vehicle of Bilastine Ophthalmic Solution; Treatment Difference (95% CI): Ketotifen Ophthalmic Solution 0.025% (Zaditen) arm minus Vehicle of Bilastine Ophthalmic Solution arm at Visit 5 (including all time points); Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.140, 95% CI 2-sided [-1.413 to -0.868]
Statistical Analysis 4: Comparison: Bilastine Ophthalmic Solution 0.6% vs Ketotifen Ophthalmic Solution 0.025% (Zaditen); Treatment Difference (one-sided, 97.5% CI): Bilastine Ophthalmic Solution 0.6% arm minus Ketotiphen Ophthalmic Solution 0.025% (Zaditen) arm at Visit 5, 3 minutes Post-CAC (non-inferiority test); Test type: Non-Inferiority — Non-inferiority margin of 0.40; p = 0.0007, ANCOVA; Mean Difference (Final Values) = 0.009, 97.5% CI 1-sided [upper limit 0.235]
Statistical Analysis 5: Comparison: Bilastine Ophthalmic Solution 0.6% vs Ketotifen Ophthalmic Solution 0.025% (Zaditen); Treatment Difference (one-sided, 97.5% CI): Bilastine Ophthalmic Solution 0.6% arm minus Ketotiphen Ophthalmic Solution 0.025% (Zaditen) arm at Visit 5, 5 minutes Post-CAC (non-inferiority test); Test type: Non-Inferiority — Non-inferiority margin of 0.40; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -0.077, 97.5% CI 1-sided [upper limit 0.175]
Statistical Analysis 6: Comparison: Bilastine Ophthalmic Solution 0.6% vs Ketotifen Ophthalmic Solution 0.025% (Zaditen); Treatment Difference (one-sided, 97.5% CI): Bilastine Ophthalmic Solution 0.6% arm minus Ketotiphen Ophthalmic Solution 0.025% (Zaditen) arm at Visit 5, 7 minutes Post-CAC (non-inferiority test); Test type: Non-Inferiority — Non-inferiority margin of 0.40; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.159, 97.5% CI 1-sided [upper limit 0.101]

ADVERSE EVENTS:
Time Frame: Safety assessment period (Day 1 through Day 8): Adverse events were assessed at all office visits, throughout a period of 8 days.
Arm/Group | Bilastine Ophthalmic Solution 0.6% | Ketotifen Ophthalmic Solution 0.025% (Zaditen) | Vehicle of Bilastine Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/90 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/90 | 0/47
Other Adverse Events (participants affected / at risk) | 4/91 | 2/90 | 1/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bilastine Ophthalmic Solution 0.6% (N=91) | Ketotifen Ophthalmic Solution 0.025% (Zaditen) (N=90) | Vehicle of Bilastine Ophthalmic Solution (N=47)
Visual Acuty Reduced (Eye disorders) | 3 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT03479307/Prot_SAP_001.pdf